CLINICAL TRIAL: NCT00641979
Title: A Multi-center, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Assess the Efficacy, Safety, and Functionality of a New Nasal Device With Reformulated Rhinocort Aqua (Budesonide) Versus the Current Product and Versus Placebo in Subjects With Seasonal Allergic Rhinitis (SAR).
Brief Title: New Nasal Applicator / New Formulation - User Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SD-005-0698; D5360C00698
Record Dates: First submitted 2008-03-18; First posted 2008-03-24 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Allergic rhinitis; Nasal symptoms; Congestion; Rhinorrhea; Sneeze; budesonide; Rhinocort AQUA
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic; Rhinorrhea; Sneezing | interventions — Budesonide

ARMS (2):
- 1 (Experimental): Rhinocort
  Interventions: Drug: budesonide; Device: Budesonide
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: budesonide — Current product
  Other Names: Rhinocort AQUA
  Arms: 1
Device: Budesonide — New type device
  Other Names: Rhinocort Aqua
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to compare the efficacy of once daily dosing with Rhinocort Aqua (new formulation) against Rhinocort Aqua (current formulation) and placebo in reliving the symptoms of seasonal allergic rhinitis (SAR).

ELIGIBILITY:
Inclusion Criteria:

* In the opinion of the investigator, is a candidate for treatment with nasal steroids based on a history of either a) inadequate control of symptoms with antihistamines, decongestants and/or immunotherapy, or b) prior successful treatment with nasal steroids.
* A documented history of at least one year of seasonal allergic rhinitis.
* A positive response to a skin prick test for grass allergens that must be present in the subject's environment throughout the study.

Exclusion Criteria:

* Primary or secondary adrenal insufficiency
* Nasal candidiasis, rhinitis medicamentosa, acute or chronic sinusitis, influenza, upper respiratory tract infection or structural abnormalities of the nose (e.g., septal deviation, nasal polyps) symptomatic enough to cause significant nasal obstruction as judged by the investigator.
* A diagnosis of asthma requiring treatment as specified in the protocol.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2002-04; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

PRIMARY OUTCOMES:
Assessment of Total Nasal Symptom scores (Rhinorrhea, Congestion, Itching & Sneezing) | 2 weekly

SECONDARY OUTCOMES:
Durability of device | End of study
Safety assessment via adverse events and clinical measurements | 2 weekly

CONTACTS AND LOCATIONS:
Overall Officials: Shaile Shah, MD, Principal Investigator — Allergy & Asthma Consultant, NJ, USA.; Bertil Andersson, Study Director — AstraZeneca